CLINICAL TRIAL: NCT04469855
Title: Post-Marketing Surveillance (Special Use-results Surveillance) on Long-term Use With Ozempic®. A Multi-centre, Open-label, Non-interventional Post-marketing Study to Investigate the Long-term Safety and Effectiveness of Ozempic® (Semaglutide) in Japanese Patients With Type 2 Diabetes Mellitus Under Normal Clinical Practice Condition
Brief Title: Post-Marketing Surveillance (Special Use-results Surveillance) on Long-term Use With Ozempic®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9535-4347; U1111-1187-9072 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ozempic®: Japanese people with type 2 diabetes being treated in normal clinical practice conditions
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Patients will be treated with commercially available Ozempic® according to routine clinical practice at the discretion of the treating physician. The treating physician's decision to initiate treatment with Ozempic® is independent of the decision to include the patient in the study.

SUMMARY:
The purpose of this study is to assess the safety of long-term treatment with Ozempic® in patients with type 2 diabetes mellitus. People will get Ozempic® as prescribed by their doctor. People will be in this study about 3 years. People above the age of 18 will be asked to fill in the quality of life (QOL) questionnaire (the QOL questionnaire is for the assessment of the influence of diabetes treatment on people's life). There is a possibility that people's blood sample would be provided to Novo Nordisk from their doctors in case of severe allergic reaction that might be caused by Ozempic®.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Ozempic® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Patients with Diabetes Mellitus, Type 2 (T2DM) who the physician has decided to start treatment with Ozempic®.
* Male or female, no age limitation.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Patients who fall under contraindications to the label.
* Patients who are or have previously been treated with Ozempic®.
* Female who is pregnant, breast-feeding or intends to become pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese people with type 2 diabetes being treated in normal clinical practice conditions
Sampling Method: Non-Probability Sample
Enrollment: 3217 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | From baseline (day 0) to end of study (month 36)
  Count

SECONDARY OUTCOMES:
Number of serious adverse reactions (SARs) | From baseline (day 0) to end of study (month 36)
  Count
Number of adverse reactions (ARs) | From baseline (day 0) to end of study (month 36)
  Count
Number of serious adverse events (SAEs) | From baseline (day 0) to end of study (month 36)
  Count
Change in glycosylated haemoglobin A1c (HbA1c) | From baseline (day 0) to end of study (month 36)
  Percent
Change in fasting plasma glucose (FPG) | From baseline (day 0) to end of study (month 36)
  mg/dL
Change in body weight | From baseline (day 0) to end of study (month 36)
  kg
Change in patient-reported outcomes (PROs) using the Diabetes Therapy-Related QOL (DTR-QOL) questionnaire - total score | From baseline (day 0) to visit 5 (month 12)
  DTR-QOL assesses the influence of diabetes treatment on the individual health related quality of life on 4 domains: "burden on social activities and daily activities", "anxiety and dissatisfaction with treatment", "hypoglycaemia" and "satisfaction with treatment". DTR-QOL contains 29 items. The response scale used is a 7-point Likert scale (1:
  Strongly agree - 7: Strongly disagree)
Change in patient-reported outcomes (PROs) using the Diabetes Therapy-Related QOL (DTR-QOL) questionnaire - burden of social activities and daily activities | From baseline (day 0) to visit 5 (month 12)
  DTR-QOL assesses the influence of diabetes treatment on the individual health related quality of life on 4 domains: "burden on social activities and daily activities", "anxiety and dissatisfaction with treatment", "hypoglycaemia" and "satisfaction with treatment". DTR-QOL contains 29 items. The response scale used is a 7-point Likert scale (1:
  Strongly agree - 7: Strongly disagree)
Change in patient-reported outcomes (PROs) using the Diabetes Therapy-Related QOL (DTR-QOL) questionnaire - anxiety and dissatisfaction with treatment | From baseline (day 0) to visit 5 (month 12)
  DTR-QOL assesses the influence of diabetes treatment on the individual health related quality of life on 4 domains: "burden on social activities and daily activities", "anxiety and dissatisfaction with treatment", "hypoglycaemia" and "satisfaction with treatment". DTR-QOL contains 29 items. The response scale used is a 7-point Likert scale (1:
  Strongly agree - 7: Strongly disagree)
Change in patient-reported outcomes (PROs) using the Diabetes Therapy-Related QOL (DTR-QOL) questionnaire - hypoglycaemia | From baseline (day 0) to visit 5 (month 12)
  DTR-QOL assesses the influence of diabetes treatment on the individual health related quality of life on 4 domains: "burden on social activities and daily activities", "anxiety and dissatisfaction with treatment", "hypoglycaemia" and "satisfaction with treatment". DTR-QOL contains 29 items. The response scale used is a 7-point Likert scale (1:
  Strongly agree - 7: Strongly disagree)
Change in patient-reported outcomes (PROs) using the Diabetes Therapy-Related QOL (DTR-QOL) questionnaire - satisfaction with treatment | From baseline (day 0) to visit 5 (month 12)
  DTR-QOL assesses the influence of diabetes treatment on the individual health related quality of life on 4 domains: "burden on social activities and daily activities", "anxiety and dissatisfaction with treatment", "hypoglycaemia" and "satisfaction with treatment". DTR-QOL contains 29 items. The response scale used is a 7-point Likert scale (1:
  Strongly agree - 7: Strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (414):
- Japan (414):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Fukushima, Japan
  - Tsuruma Kaneshiro Diabetes Clinic_Internal medicine, Yamato-shi, Kanagawa
  - Takai Medical Clinic_Internal Medicine, Kamakura-shi, Kanagawa, Kanagawa, Japan
  - Matsuba Clinic_Internal Medicine, Kawasaki-shi, Kanagawa, Japan
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Abe Diabetes Clinic_Internal Medicine, Ōita, Oita, Japan
  - Iryo Houjin Hakuunkai Ryoya Komatsu Clinic,Internal medicine, Izumisano, Osaka, Japan
  - Asano Clinic, Kawagoe-shi, Saitama, Japan
  - Tokyo Saiseikai Central Hospitl, Internal Med, Minatoku, Tokyo, Japan
  - Ohgaku Clinic, Internal Medicine, Imizu-shi, Toyama, Japan
  - Yamauchi Family Clinic, Aichi
  - Kobayashi Naika Clinic, Aichi
  - Wakaba Clinic, Aichi
  - Miyachi Clinic, Aichi
  - Meiekihigashi Clinic, Aichi
  - Meitetsu Hospital_Endocrinology and Metabolism, Aichi
  - Kusama Minato Clinic, Aichi
  - Nagashima Naika, Aichi
  - Aikawa Minnano Shinryojo, Aichi
  - Nakai Internal Clinic, Aichi
  - Takenaka Clinic, Aichi
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Enomoto Naika, Aichi
  - Sawayaka Medical Clinic, Aichi
  - Ogawa Clinic_Aichi, Aichi
  - Inuyama Chuo General Hospital_Diabetes Internal Medicine, Aichi
  - Uenishi Internal Medicine Clinic, Aichi
  - Tosei General Hospital_Endocrinology and Metabolism, Aichi
  - Noshiro Kosei Iryo Center_Diabetes and Metabolism, Akita
  - Odate Municipal General Hospital_Endocrinology and Metabolism, Akita
  - Kitaakita Shiritsu Yonaizawa Shinryojo, Akita
  - Ohisama Clinic_Aomori, Aomori
  - Kakizaki Tonyobyo Naika Clinic, Aomori
  - Kumanomae Nishimura Naika Clinic_Internal Medicine, Arakawa-ku, Tokyo
  - Shimizu internal medicine clinic, Asahikawa-shi, Hokkaido
  - Chiba Central Medical Center, Chiba
  - Shimada Iin, Chiba
  - Ichikawaekimae Ogawa Naika, Chiba
  - Endo Naika, Chiba
  - Misaki Naika Clinic, Chiba
  - Shinkashiwa Clinic Tonyobyomirai, Chiba
  - The Jikei University Kashiwa Hospital_Diabetes and Endocrinology, Chiba
  - Tokyo Bay Urayasu Ichikawa Medical Center_Neph.& Endocrinology, Diabetes, Chiba
  - Saito Clinic, Chiba
  - Toyo Clinic, Chiba
  - Chiba Cerebral and Cardiovascular Center, Chiba
  - Kimitsu Chuo Hospital_Diabetology and Endocrinology, Chiba
  - Matsunaga Iin, Chiba
  - Gengendo Kimitsu Hospital_Diabetes and Endocrinology, Chiba
  - Akaicho Clinic, Chiba-shi, Chiba
  - Mizuno Clinic, Chichibu
  - Hasegawa Medicine Clinic, Internal medicine, Chitose, Hokkaido
  - Soyokaze CardioVascular Medicine and Diabetes Care, Ehime
  - Mikannohana Clinic, Ehime
  - Ehime Medical Center, Ehime
  - Yoshino Internal Medicine, Ehime
  - Matsuyama Daiichi Hospital_Diabetes Internal Medicine, Ehime
  - Saiseikai Matsuyama Hospital_Internal Medicine, Ehime
  - Ehime Prefectural Niihama Hp._Internal Medicine, Ehime
  - Jyuzen General Hospital_Internal Medicine, Ehime
  - Hoshasen Daiichi Byoin_Internal Medicine, Ehime
  - Uwajima City Hospital_Endocrinology and Diabetes, Ehime
  - Shikoku Central Hospital_Internal Medicine, Ehime
  - Fukui Chuoh Clinic, Fukui
  - Fukui Prefecture Saiseikai Hospital, Internal Medicine, Fukui-shi, Fukui
  - Kyushu Rosai Hospital_Diabetes and Metabolism, Fukuoka
  - Kuroki Hiro Clinic, Fukuoka
  - Hatanaka Naika Clinic, Fukuoka
  - Minezaki Naika Clinic, Fukuoka
  - Chiyo Clinic, Fukuoka
  - Hayashida Internal Medicine Clinic, Fukuoka
  - Okabe Hospital_Internal Medicine, Fukuoka
  - Fukutsu Naika Clinic, Fukuoka
  - Okada Naika Clinic, Fukuoka
  - Tojitama Thyroid and Diabetes Clinic, Fukuoka
  - Clinic Masae Minami, Fukuoka
  - Iino Naika, Fukuoka
  - Kikuchi Naika Iin Maebaru, Fukuoka
  - Iizuka Kaho Hospital_Internal Medicine, Fukuoka
  - Kuwano Naika Shonika Iin, Fukuoka
  - Ishibashi Iin, Fukuoka
  - Chikugo Shiritsu Byoin_Endocrinology and Metabolism, Fukuoka
  - Himeno Hospital, Fukuoka
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Iwashina Clinic, Fukushima
  - Aizu Clinic, Fukushima
  - Taneda Clinic, Fukushima
  - Tani Naika Clinic, Internal medicine and diabets, Fukushima-shi, Fukushima
  - Yamauchi Hospital_Internal Medicine, Gifu
  - Keyaki Clinic, Gifu
  - Kitada Internal Medicine Clinic, Gifu
  - Matsunami General Hospital_Diabetes and Endocrinology, Gifu
  - Asano Naika, Gifu
  - Ogawa Clinic_Gifu, Gifu
  - Gifu University Hospital,The Third Dep of Internal Medicine, Gifu-shi, Gifu
  - Shimizu Naika, Gunma
  - Kawada Clinic, Gunma
  - Goga Internal Medicine Nire Clinic, Gunma
  - Takekawa clinic, Internal Medicine, Higashiosaka-shi, Osaka
  - Sato Family Clinic, Hiroshima
  - Tanabe Clinic, Hiroshima
  - Murakami Memorial Hospital_Diabetes Internal Medicine, Hiroshima
  - Hiroshima Red Cross & Atomic-b_Endocrinology and Metabolism, Hiroshima
  - Hisayasu Iin, Hiroshima
  - Higashihiroshima Medical Center, Hiroshima
  - Takasawa Diabetes Clinic, Hokkaido
  - Nakagaki Primary Care Clinic, Hokkaido
  - Ohata Naika Junkanki Clinic, Hokkaido
  - Sapporo Tonyobyo Kojosen Clinic Asty45, Hokkaido
  - Okamoto Naika Clinic_Hokkaido, Hokkaido
  - Sapporo Tonyobyo Kojosen Clinic, Hokkaido
  - Hokkaido Medical Center, Hokkaido
  - Ito Hiroshi Naika Tonyobyonaika Clinic, Hokkaido
  - Sapporo Yamahana Internal Medicine & Diabetes Clinic, Hokkaido
  - Yoshimura Tonyobyo Clinic, Hokkaido
  - Japanese Red Cross Asahikawa Hospital, Hokkaido
  - Kagetsu Clinic, Hokkaido
  - Yamagata Naika Clinic, Hokkaido
  - Honjo Naika Clinic, Hokkaido
  - Owari Cardiovascular Diabetes Medicine Clinic, Hosu-gun, Ishikawa
  - Takabe Diabetes Clinic, Hyogogoken
  - Shinkobe Okada Clinic, Hyōgo
  - Kaisei Clinic, Hyōgo
  - Hishikawa Naika Clinic, Hyōgo
  - Konan Medical Center_Diabetes and Endocrinology, Hyōgo
  - Sumiyoshigawa Byoin_Diabetes and Internal Medicine, Hyōgo
  - Ashiya Municipal Hospital_Diabetes and Endocrinology, Hyōgo
  - Yamasaki Family Clinic, Hyōgo
  - Mitsuru Clinic, Hyōgo
  - Taniguchi Medical Clinic, Hyōgo
  - Azuma Diabetes Clinic, Hyōgo
  - Nakayamadera Imai Clinic, Hyōgo
  - Tsukazaki Memorial Hospital_Internal Medicine, Hyōgo
  - Himeji St.Mary's Hospital_Gastroenterology - Hepatology, Hyōgo
  - Fukatsu Naika Shinryojo, Hyōgo
  - Yokota Medical Clinic, Hyōgo
  - Akashi Medical Center, Hyōgo
  - Tateya Clinic, Hyōgo
  - Hirai Naika Clinic, Hyōgo
  - Ono Hospital_Internal Medicine, Hyōgo
  - Hyogo Prefectural Kakogawa Medical Center_Diabetes and Endocrinology, Hyōgo
  - Obata Naika Tonyobyo Clinic, Hyōgo
  - Ako City Hospital_Internal Medicine, Hyōgo
  - Tsuchiura Shinryo Kenshin Center, Ibaraki
  - Tokyo Medical University Ibaraki Medical Center_Metabolism and Endocrinology, Ibaraki
  - Iwaki Internal Medicine Clinic, Ibaraki
  - Itabashi Diabetes and Dermatology Medical Clinic, Ibaraki
  - Tomobe Central Clinic, Ibaraki
  - Mito Kyodo General Hospital_Diabetes and Endocrinology, Ibaraki
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Maeda Hospital_Internal Medicine, Ibaraki
  - Ohta Clinic, Internal Medicine, Iruma-shi, Saitama
  - Isobe Tounyoubyou Naika Clinic, Ishikawa
  - Kanazawa Medical University Hospital_Endocrinology and Metabolism, Ishikawa
  - Kagawa Prefectural Central Hospital_Diabetes and Endocrinology, Kagawa
  - Akiyama Clinic, Kagawa
  - Takahashi Seikeigeka Iin, Kagawa
  - Osugi Neurosurgical Clinic, Kagawa
  - Iwamoto Internal Medicine Clinic_Diabetes Internal Medicine, Kagawa
  - Tsuda Shinryojo, Kagawa
  - Uenomachi Kajiya Clinic, Kagoshima
  - Keiai Clinic, Kagoshima
  - Fukuda Iin, Kagoshima
  - Sonoda Clinic, Kagoshima
  - Wakamatsu Kinen Byoin_Internal Medicine, Kagoshima
  - Shimozono Clinic, Kagoshima
  - Aira Tonyobyo Kojosen Naika Clinic, Kagoshima
  - Tempozan Clinic of Internal Medicine, Kagoshima-shi, Kagoshima
  - Sun Marco Clinic, Kanagawa
  - Nakahara Medical Clinic, Kanagawa
  - Teikyo Univ.HP, Mizonokuchi_Fourth Internal Medicine, Kanagawa
  - Kubota Clinic, Kanagawa
  - Nishikawa Clinic, Kanagawa
  - Tsunashima East Internal med & Diabetes, Kanagawa
  - Yokohama City Minato Red Cross Hospital_Endocrinology, Kanagawa
  - H.E.C Science Clinic, Kanagawa
  - Kikuchi Naika Clinic_Kanagawa, Kanagawa
  - Yokohama Minami Kyousai Hospital_Cardiology, Kanagawa
  - Tagawa Naika Iin, Kanagawa
  - Suzuki Diabetes Clinic, Kanagawa
  - Yokohama Medical Center_Diabetes and Endocrinology, Kanagawa
  - Shonan Takai Clinic_Internal Medicine, Kanagawa
  - Odawara Municipal Hospital_Diabetes and Endocrinology, Kanagawa
  - Sawa Internal Medicine and Diabetes Clinic, Kanagawa
  - Internal Medicine Clinic Kobayashi, Kanagawa
  - Higashirinkan Kaneshiro Diabetes Clinic, Kanagawa
  - Chigasaki Municipal Hospital_Endocrinology and Metabolism, Kanagawa
  - Hiratsuka Kyosai Hospital_Endocrinology and Metabolism, Kanagawa
  - Kyourindo Clinic, Kanagawa
  - Seichi Clinic, Kanagawa
  - Tokai University Hospital_Cardiology, Kanagawa
  - Hotaruno hakuyukai Medical Corporation of Japan, Kisarazu-shi, Chiba
  - Kobe University Hospital_Diabetes and Endocrinology, Kobe, Hyogo
  - Ueta Iin, Kochi
  - Kikuchi Naika Clinic, Kokuryō
  - Ringo no Hana Clinic, Kokuryō
  - Morimura Clinic, Kokuryō
  - Arai Shinryojo, Kokuryō
  - Koshigaya Laketown Clinic, Koshigaya-shi,Saitama
  - Tamana Central Hospital_Diabetes and Endocrinology, Kumamoto
  - Minamata City General Hospital & Medical Center_Metabolism, Kumamoto
  - Jujo Takeda Rehabilitation Hospital_Diabetes Internal Medicine, Kyoto
  - Kyoto Goshominami Harashima Clinic, Kyoto
  - Kamiuchi Naika Clinic, Kyoto
  - Toyoda Medical Clinic, Kyoto
  - Mata Clinic, Kyoto
  - Oishi Naika Clinic, Kyoto
  - Koide Iin, Kyoto
  - Ayabe City Hospital_Endocrinology and Diabetes, Kyoto
  - Mie Chuo Medical Center_Internal Medicine, Mie
  - Mie University Hospital_Mie, Mie
  - MG Clinic, Mie
  - Japanese Red Cross Ise Hospital_Diabetes and Metabolism, Mie
  - Kanno Naika_Internal Medicine, Mitaka-shi, Tokyo
  - Miura Central Clinic, Miura-shi, Kanagawa
  - Shirai Healthcare Clinic Izumi-chuo, Miyagi
  - Suzuki Kenichi Naika Clinic, Miyagi
  - Yoshizumi Clinic Diabetes and Endocrinology, Miyagi
  - Morita Iin, Miyagi
  - Koga General Hospital_Internal Medicine, Miyazaki
  - Mitsukawa Naika Iin, Miyazaki
  - Nichinan Chubu Hospital_Internal Medicine, Miyazaki
  - Sumi Byoin_Internal Medicine, Miyazaki
  - Ato internal medicine clinic, internal medicine, Muroran-shi, Hokkaido
  - Asama General Hospital_Diabetology, Nagano
  - Houden Clinic, Nagano
  - Shinshu Ueda Medical Center_Diabetes and Endocrinology, Nagano
  - Iida Municipal Hospital_Diabetes and Metabolism, Nagano
  - Kenwakai Hospital_Dialysis center, Nagano
  - Ina Central Hospital_Internal Medicine, Nagano
  - Saiseikai Nagasaki Hospital_Endocrinology and Diabetes, Nagasaki
  - Yuzu Clinic, Nagasaki
  - Onitsuka Naika Shokakika, Nagasaki
  - Miyazaki Naika, Nagasaki
  - Tetsuo Naika Iin, Nagasaki
  - Japanese Red Cross Nagasaki Genbaku Hospital_Metabolism and Endocrinology, Nagasaki
  - Nakamura Iin, Nagasaki
  - Sasebo City General Hospital_Diabetes and Endocrinology, Nagasaki
  - Harada Tonyobyo Jin Naika Clinic, Nara
  - Hikari Clinic, Nara
  - Imamura Tonyobyo Naika Tsuda Geka Shinryojo, Nara
  - Furuya Clinic, Nara
  - Okamoto Internal Medicine and Pediatrics Clinic, Nara
  - Mashitani Naika Clinic, Nara
  - Ikenaka Naika Clinic, Nara
  - Seiwadai Clinic, Nara
  - Enomoto Clinic, Nara
  - Minagawa Clinic Internal Medicine, Niigata
  - Takahashi Iin, Niigata
  - Uchiyama Iin, Niigata
  - Niigata Prefectural Sakamachi Hospital_Internal Medicine, Niigata
  - Saiseikai Niigata Hospital_Metabolism and Endocrinology, Niigata-shi, Niigata
  - Hyogo College Hospital_Diabetes and Endocrinology, Nishinomiya-shi, Hyogo
  - Kaneko Gastroenterologist Internal Medicine, Numakunai
  - Abies Kanno Clinic, Numakunai
  - Kitakamiekimae Naika Clinic, Numakunai
  - Iwate Medical University Hospital_Diabetes and Metabolism, Numakunai
  - Okayama University Hospital_General Medicine, Okayama
  - Obata Medical Clinic, Okayama
  - Shigei Byoin_Internal Medicine, Okayama
  - Kojima Marine Clinic, Okayama
  - Kasaoka Daiichi Hospital_Internal Medicine, Okayama
  - Okayama Medical Center_Cardiology, Okayama-shi, Okayama
  - Tokuyama Clinic, Okinawa
  - Shuri Jokamachi Clinic, Okinawa
  - Chibana Clinic, Okinawa
  - Sunagawa Medical Clinic, Okinawa
  - Taiyono Clinic, Okinawa
  - Tanaka Naika, Osaka
  - Nishimura Clinic, Osaka
  - Manabe Iin, Osaka
  - Osaka City General Hospital_Endocrinology and Diabetes Mellitus, Osaka
  - Yasuda Diabetes Clinic, Osaka
  - Osaka National Hospital_Diabetes Internal Medicine, Osaka
  - Kosugi Medical Clinic, Osaka
  - Osaka Police Hospital_Diabetes and Endocrinology, Osaka
  - Osaka City University Hospital_Metabolism and Endocrinology, Osaka
  - Matsumoto Clinic, Osaka
  - Kansai Electric Power Hospital_Center for Diabetes, Osaka
  - Ichiyoshi Iin, Osaka
  - Osaka General Medical Center_Cardiology, Osaka
  - Jo's Medical Clinic, Osaka
  - Minamitani Clinic, Osaka
  - Nakanishi Clinic, Osaka
  - Mori Clinic, Osaka
  - Maeda Clinic, Osaka
  - Masuda Clinic, Osaka
  - Sawaki Internal Medicine And Diabetes Clinic, Osaka
  - Hokusetsu General Hospital_Diabetes and Endocrinology, Osaka
  - Matsushita Memorial Hospital_Diabetes and Endocrinology, Osaka
  - Tesseikai Noshinkeigeka Byoin_Cardiology, Osaka
  - Iwasaki Naika Clinic, Osaka
  - Ogawa Clinic, Osaka
  - Matsuda Gastroenterology and Diabetes Clinic, Osaka
  - Jonin Ueda Clinic, Osaka
  - Tamai Hospital_Diabetes Internal Medicine, Osaka
  - Minami Sakai Hospital_Internal Medicine, Osaka
  - Bellland Sogo Byoin_Endocrinology and Metabolism, Osaka
  - Fukuda Clinic, Internal Medicine, Osaka-shi, Osaka
  - Yodogawa Christian Hospital, Osaka-shi, Osaka
  - Saiseikai Noe Hospital, Osaka-shi, Osaka
  - Osaki citizen hospital_Diabetes and metabolic disease, Osaki-shi, Miyagi
  - Iryo Houjin Shadan Sosyu-kai SATO MEDICAL CLINIC, Ota-ku, Tokyo
  - Shin Clinic, Ota-ku, Tokyo
  - Oita Prefectural Hospital_Endocrinology and Metabolism, Ōita
  - Kayashima Clinic, Ōita
  - Cosmos Byoin_Internal Medicine, Ōita
  - Takada Chuo Byoin_Diabetes Internal Medicine, Ōita
  - Okamoto Clinic for Diabetes and Endocrinology, Ōita
  - Nagomitoiyashino Clinic, Saga
  - Noda Kousei Clinic, Saga
  - Noguchi Internal Clinic, Saga
  - Seki Clinic, Saga
  - Karatsu Redcross Hospital_Diabetes Internal Medicine, Saga
  - Saga National Hospital_Internal Medicine, Saga
  - Saitama Medical Center_Diabetes and Endocrinology, Saitama
  - Tanaka Clinic_Saitama, Saitama
  - Nakayama Clinic, Saitama
  - Ishizuka Medical Clinic, Saitama
  - Yokota Iin, Saitama
  - Kanazawa Clinic, Saitama
  - Josai Naika Clinic, Saitama
  - Negishi Naika Taisha Clinic, Saitama
  - Mami clinic of internal medicine, Saitama
  - Imaki Clinic, Saitama
  - Arafune Clinic, Saitama
  - Matsudakai Tsurugaya Clinic, Internal medicine, Sendai-shi, Miyagi
  - Tonyobyo Clinic Katata, Shiga
  - Kaneda Iin, Shiga
  - Omihachiman Community Medical Center_Metabolism and Endocrinology, Shiga
  - Nagahama City Hospital_Nephrology and Metabolism, Shiga
  - Nabika Naika Clinic, Shimane
  - Kanazawa Diabetes & Osteoporosis Clinic, Shimane
  - Takase Naika, Shimane
  - Sekiminatokinenkai Green Clinic, Shimotsuga-gun, Tochigi
  - Wakakusa Clinic, Shimotsuke-shi, Tochigi
  - Center Hospital of the National Center for Global Health and Medicine_Cardiovascular Medicine, Shinjuku-ku, Tokyo
  - Medical corporation group lifestyle Tomonaga clinic_Internal Medicine, Shinjyuku-ku Tokyo
  - Aso Clinic, Shizuoka
  - Mochizuki Naika Iin, Shizuoka
  - Yata Ikeda Iin, Shizuoka
  - Goto Clinic, Shizuoka
  - Japan Red Cross Shizuoka Hospital_Diabetes and Endocrinology, Shizuoka
  - Kikuchi Medical Clinic, Shizuoka
  - Hamamatsu-kita-Hospital_Internal Medicine, Shizuoka
  - Hamamatsu Medical Center, Shizuoka
  - Shizuoka city Shizuoka Hospital_Endocrinology and Metabolism, Shizuoka-city, Shizuoka
  - Soka Sugiura Internal Medicine Clinic, Soka-shi, Saitama
  - Nagano Prefectural Shinshu Medical Center., Suzaka-shi ,Nagano
  - Higashi Diabetes and Cardiovascular Clinic, Internal, Tamana-shi, Kumamoto
  - Kawakami Hospital_Internal Medicine, Tochigi
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Nagasaki Hospital_Internal Medicine, Tochigi
  - Saino Clinic, Tokorozawa-shi,Saitama
  - Ooshima Clinic, Tokushima
  - Iwaki Clinic_Diabetes Internal Medicine, Tokushima
  - Tamaki Aozora Byoin_Diabetes and Endocrinology, Tokushima
  - Mitsui Memorial Hospital_Diabetes and Metabolism, Tokyo
  - Kudanzaka Hospital_Internal Medicine, Tokyo
  - Hamacho Center Bldg. Clinic, Tokyo
  - Ginza Yasue Clinic, Tokyo
  - Hosokawa Clinic, Tokyo
  - The Jikei University Hospital Dept of Diabetes, Metabolic, Tokyo
  - Shirokanedai Ogawa Clinic, Tokyo
  - Kitasato Institute Hospital_Diabetes Center, Tokyo
  - Ueno Asakusa Street Clinic, Tokyo
  - Kyowa Iin, Tokyo
  - Kato Medical Clinic, Tokyo
  - Mikawashima Tower Clinic, Tokyo
  - Suzuki Diabetes Clinic_Tokyo, Tokyo
  - The Jikei University Katsushika Iryo Center_Diabetes and Endocrinology, Tokyo
  - Seikodo Clinic, Tokyo
  - Asoka Hospital_Internal Medicine, Tokyo
  - Okamoto Naika Clinic, Tokyo
  - Cancer Institute Ariake Hosp._Diabetes and Metabolism, Tokyo
  - Togoshi Perk Clinic, Tokyo
  - Makita General Hospital_Diabetes Internal Medicine, Tokyo
  - Toho University Omori Medical Center_Diab Metab Endo, Tokyo
  - Kamata Diabetes Clinic, Tokyo
  - Takeuchi Naika Shonika Iin, Tokyo
  - Matsuura Clinic, Tokyo
  - Mishuku Hospital, Tokyo
  - Kokubo Clinic, Tokyo
  - Shimokitazawa Hospital_Diabetes Center, Tokyo
  - Ohkubo Hospital_Endocrinology and Metabolism, Tokyo
  - Tokyo General Hospital_Diabetes and Metabolism, Tokyo
  - Ekimae Tsunoda Clinic, Tokyo
  - Nerima General Hospital_Internal Medicine, Tokyo
  - KAWASAKI internal medicine clinic & Diabetic, Tokyo
  - Hoya Iin, Tokyo
  - Clinic Mirai Kunitachi, Tokyo
  - Clinic Mirai Tachikawa, Tokyo
  - Hachioji Diabetes Clinic, Tokyo
  - Tokyo Medical Univ. Hachioji_Diabetes and Endocrinology, Tokyo
  - Sato Juichi Clinic, Tokyo
  - Ome Municipal General Hospital_Endocrinology and Metabolism, Tokyo
  - Higashikurume Ekimae Clinic, Tokyo
  - Tamacenter Clinic Mirai, Tokyo
  - Tanaka Clinic, Tomigusuku-shi, Okinawa
  - Satoni Denen Clinic, Tottori
  - Tottori University Hospital_Cardiovascular Medicine, Tottori
  - Shinseikai Toyama Hospital_Diabetes Center, Toyama
  - Toyama University Hosp., Dept. of Diabetes, Metabo.& Endoc., Toyama-shi, Toyama
  - Senrichuo Ekimae Clinic, Toyonaka-shi, Osaka
  - Japanese Red Cross Wakayama Medical Center_Diabetology and Endocrinology, Wakayama
  - Tohoku Central Hospital_Diabetes Internal Medicine, Yamagata
  - Kochi Iin, Yamagata
  - Iwasaki Naika Iin, Yamaguchi
  - Okino Naika Tonyobyo Clinic, Yamaguchi
  - Yamaguchi Rosai Hospital_Diabetes and Endocrinology, Yamaguchi
  - Nakazato Medical Clinic, Yamanashi
  - Nagata Hospital, Yanagawa-shi, Fukuoka
  - Yokohama Rosai Hospital, Yokohama, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com